CLINICAL TRIAL: NCT01936506
Title: Cognitive Training for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 10-0645
Record Dates: First submitted 2013-08-29; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Major Depressive Disorder
Keywords: Cognitive training; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training A (Experimental): emotional memory training exercise
  Interventions: Behavioral: Cognitive Training A
- Cognitive Training B (Active Comparator): memory training exercise
  Interventions: Behavioral: Cognitive Training B

INTERVENTIONS:
Behavioral: Cognitive Training A
  Arms: Cognitive Training A
Behavioral: Cognitive Training B
  Arms: Cognitive Training B

SUMMARY:
This study is evaluating the effects of two brain training exercises on: memory, cognitive processing and depression symptoms.

DETAILED DESCRIPTION:
There is an urgent public health need to develop more effective and well tolerated treatments for patients with major depressive disorder (MDD); cognitive training interventions aiming to modify cognitive and affective processing abnormalities underlying MDD represent a promising new strategy. This research project translates a well established cognitive bias in major depressive disorder (MDD), working memory bias, into a novel intervention target. In a double-blind, randomized, controlled study, MDD participants undergo 4 weeks of cognitive training sessions, with two sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Primary, current Axis I diagnosis of Major Depressive Disorder according to DSM-IV criteria and Ham-D-17 score between 16-27
* Age 18-55
* Able to give informed consent

Exclusion Criteria:

* A history of drug or alcohol abuse or dependence (DSM-IV criteria) within 6 months
* Visual impairment that would affect the ability to observe the computerized presentation of faces.
* Motor impairment that would affect the ability to provide a response by quickly pressing a button.
* Lifetime history of Bipolar spectrum disorders or schizophrenia spectrum disorders.
* Primary, current Axis I diagnosis other than Major Depressive Disorder
* Primary, current Axis II personality disorder.
* Currently attending a cognitive-behavioral psychotherapy regimen
* Acute suicidal or homicidal risk (evidenced by suicidal or homicidal attempt within 6 months of screening)
* Pregnancy in women.

Subjects must exhibit no or only moderate alcohol use. Subjects with current excessive use of alcohol (> 8 ounces/day for men and > 6 ounces/day for women) are ineligible for participation, as such drug use could confound the results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
change in Hamilton Depression Rating Scale (Ham-D) | baseline and week 4
  Change in depression symptom severity at week 4 compared as to baseline

SECONDARY OUTCOMES:
change in Self-referential Information Processing Task | baseline and week 4
  change in Negative Affective Bias at week 4 as compared to baseline
change in Working Memory | baseline and week 4
  change in Neurocognition at week 4 as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Iacoviello, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States